CLINICAL TRIAL: NCT06601374
Title: Characteristics and Outcomes of Patients With Pregnancy Related Acute Kidney Injury in Assiut University Hospitals: a Single-center Study
Brief Title: Patient Presented With AKI Related to Pregnancy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Saber Mohamed Ali, MBBCH , principal investigator, Assiut University
Other Study IDs: Pregnancy related AKI
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Kidney Injury
Keywords: AKI related to pregnancy; AKI; PRAKI; Pregnancy related AKI
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to identify characteristics of patient with PR AKI treated in Assiut university hospital

Secondary outcomes:

1. Assessment of pregnancy related AKI maternal outcome (complete recovery , partial recovery or progress to ESRD) within 3 months duration
2. To identify predictors of unfavorable outcome of patient with pregnancy related AKI

DETAILED DESCRIPTION:
Acute kidney Injury (AKI) is a syndrome which is characterized by an rapid deterioration of the kidney function , manifested by increase in serum creatinine level with or without reduced urine output and linked to high rate of morbidity and mortality .AKI is considered a major public health problem despite much improvmnent in heakth care and especially, most of them (about 85 %) in developing countries with low resources.Pregnancy related AKI ( PR -AKI ) is a major obstetric complication which may cause termination of pregnancy (TOP ), Intensive care unit ( ICU ) admission , need for dialysiy , both maternal and perinatal morbidity and mortality with maternal mortality rang from 9% to 55 % .

PR-AKI has a major risk factors include preeclampsia which is the most common cause (15-20%) , hyperemesis gravidarum , acute fatty liver of pregnancy and placental abruption , puerperal sepsis and septic abortion .The maternal outcome of pregnancy related AKI include complete recovery with return of serum creatinine to normal (> 1.4 mg /dl ) about (40-75% ), partial recovery(4-9% require dialysis about 4 months after delivery) , progress to End stage renal disease (1.5 - 2.5 %) or maternal mortality . The maternal mortality rate (MMR) increases with increasing severity of pregnancy-related complications and can range from 13 to 24% in developing countries due to PR-AKI .

Timely identification of patients and management of underlying conditions is considered the cornerstone to improve maternal outcome.

ELIGIBILITY:
Inclusion Criteria:

* Women (>18 years) who developed AKI with or without need for dialysis treatment during pregnancy, childbirth , post abortion period and /or puerperium
* AKI as defined by KDIGO definition as follows:

  1. Increase in serum creatinine > 0.3 mg/dl within 48
  2. Increase in serum creatinine > 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days.
  3. urine volume of < .5 ml / kg / hours

Exclusion Criteria:

* Patients with preexisting kidney disease before pregnancy
* Patients with AKI not related to pregnancy.
* Patients with uncertain history for incident time of AKI.
* Patients refuse to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female presented with AKI related to pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The occurance of renal recovery | After the insult and up to the subsequent 3 month duration
  The occurance of renal recovery measured by serum creatinine , eGFR , urinary proteins and need for dialysis after the insult and up to the subsequent 3 month duration

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Saber, MBBCH, Principal Investigator — Assiut university _ faculty of medicine; Mahmoud Ali, MBBCH, Study Director — Assiut university _ faculty of medicine